CLINICAL TRIAL: NCT00209079
Title: Phase II Trial of Gleevec (Imatinib Mesylate) and Taxotere (Docetaxel) as a Combined Regimen for Advanced Gastric Adenocarcinoma
Brief Title: Phase II Trial of Gleevec and Taxotere as a Combined Regimen for Advanced Gastric Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated 4/17/07. Drug sponsor withdrew.
Sponsor: Emory University (Other)
Collaborators: Novartis (Industry)
Responsible Party: John Kauh, MD, Winship Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0804-2004
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2007-12-31 (Estimated); Status verified 2007-09

CONDITIONS: Gastric Adenocarcinoma
Keywords: Gastric Adenocarcinoma
MeSH Terms: interventions — Imatinib Mesylate; Docetaxel; Mesylates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator)
  Interventions: Drug: Gleevec, Taxotere

INTERVENTIONS:
Drug: Gleevec, Taxotere — Gleevec taken 4 times daily, 100 mg per tablet. Taxotere intravenously once a week for two weeks.
  Other Names: Imatinib, Mesylate, Docetaxel

SUMMARY:
The purpose of this trial is to test the combination of Gleevec® (also known as imatinib mesylate) and Taxotere (also known as docetaxel) in patients with incurable stomach cancer. This study is being performed to see if the combination of Gleevec and Taxotere is an effective treatment for incurable stomach cancer with minimal side effects.

DETAILED DESCRIPTION:
The purpose of this trial is to test the combination of Gleevec® (also known as imatinib mesylate) and Taxotere (also known as docetaxel) in patients with incurable stomach cancer. Gleevec is a pill form of chemotherapy and is indicated for the treatment of adult patients with chronic myeloid leukemia (CML) and gastrointestinal stromal tumors (GIST). It is considered experimental for the treatment of stomach cancer. Taxotere (docetaxel) is a chemotherapy which is injected into the vein. It is approved for breast and lung cancer but has been shown to shrink many different types of tumors. Taxotere has been shown to shrink stomach cancer in about 20% - 30% of patients treated with Taxotere only. This study is being performed to see if the combination of Gleevec and Taxotere is an effective treatment for incurable stomach cancer with minimal side effects.

Treatment on this study consists of two drugs, Gleevec® and Taxotere. Patients will be take four tablets of Gleevec® daily throughout the study. After one week of Gleevec®, patients will then begin receiving doses of Taxotere intravenously once a week for two weeks in a row followed by one week without Taxotere.

ELIGIBILITY:
Inclusion Criteria:

* This study is for patients with histologically confirmed unresectable gastric adenocarcinoma and who have not received any chemotherapy other than 5-FU for adjuvant therapy either alone or in conjunction with radiation.

Exclusion Criteria:

* Patients may not have received any chemotherapy agents other than 5-FU.
* Patients may not have received 5-FU for for therapy for metastatic gastric cancer.
* Patients must be more than 5 years free of another primary malignancy except: if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
* Patients must not have Grade III/IV cardiac problems, or any severe and/or uncontrolled medical disease (i.e. uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
* Patient must not have had previously received radiotherapy to >/= 25% of the bone marrow, or have had major surgery within 2 weeks prior to study entry
* Final eligibility for a clinical trial is determined by the health professionals conducting the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2004-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Determine if combination of Gleevec and Taxotere is effective treatment for incurable stomach cancer. | 3 months

SECONDARY OUTCOMES:
Determine toxicity of combination of Gleevec and Taxotere. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: John Kauh, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States